CLINICAL TRIAL: NCT01801033
Title: Effects of Pharmacologic Block of Type-1 Deiodinase on Thyroid Hormone Action and on the Circulating Levels of T3 in Hypothyroid Patients
Brief Title: Effects of Thyroid Hormone Enzyme Blocking on Hypothyroidism
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130058; 13-DK-0058
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2013-11-29

CONDITIONS: Hypothyroidism; Thyroidectomy
Keywords: Trioodothyronine (T3); Thyroid Hormone Action; Deiodinases; Hypothyroid; Propylthiouracil (PTU)
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Hypothyroidism is a condition caused by the loss of function of the thyroid gland. The thyroid gland produces two hormones, T4 and T3. These hormones control the metabolism and function of many organs. Lack of energy, depression, and constipation are common symptoms of hypothyroidism. T4 is converted into T3, the active form of thyroid hormone, by two enzymes called deiodinases. People with hypothyroidism are treated with a synthetic T4 hormone, which the enzymes convert to T3. This treatment is usually effective, but some people continue to have symptoms even after treatment. Some researchers think that this may be caused by a problem with the enzymes that convert T4 into T3. They want to look at how the enzymes regulate the levels of T4 and T3 in the blood. They will do so by using a drug that blocks the action of one of the two enzymes.

Objectives:

- To look at how thyroid hormone enzyme blocking affects hypothyroidism treatment medication.

Eligibility:

- Individuals at least 18 years of age who have hypothyroidism and are on thyroid hormone replacement therapy.

Design:

* The study consists of one screening visit, 9 days of inpatient hospital admission, and a follow-up visit 2 weeks after discharge.
* Participants will be screened with a physical exam and medical history. They will provide blood samples.
* Participants will receive balanced-diet meals to take home for the 2 days before they enter the hospital. They will continue this diet while in the hospital.
* During the inpatient stay, participants will be monitored with regular blood tests. They will have the following procedures:
* Continued thyroid hormone replacement for all 9 days.
* Drug to block thyroid enzyme for 7 days.
* Metabolism test, with room temperature changes, on days 1, 2, 5, 8, and 9.
* Measurements of body fat on days 2, 5, and 8.
* Blood glucose tests on days 1 and 9.
* Muscle contraction tests on days 1, 2, 4, 5, 8, and 9.
* Heart imaging studies on days 2, 5, and 8.
* Optional skeletal muscle and fat tissue biopsies on days 1 and 9.
* There will be a follow-up visit 2 weeks after leaving the hospital. Participants will have a final physical exam and provide blood samples.

DETAILED DESCRIPTION:
Thyroid hormone action is an important regulator of the metabolism and the function of many organs. The active form of thyroid hormone is T3, and its blood and tissue levels are the result of the secretion of T3 and its precursor, thyroxine (T4), from the thyroid gland, of the peripheral conversion of T4 into T3, and of the degradation of these hormones. In hypothyroid patients (particularly patients who underwent total thyroidectomy), the levels of T3 are entirely dependent on the exogenously administered T4 (Levothyroxine, L-T4) which is converted to T3 or to the inactive form, rT3, by enzymes called deiodinases. This complex system has only been partially studied in humans and very little is known about the correlation between circulating levels of T3 and end-organ target tissue thyroid hormone action.

The aim of this protocol is to characterize the contribution of the two activating deiodinases (type-1 and type-2) to the blood levels and biological effects of T3. To achieve this goal we intend to study hypothyroid patients treated with adequate replacement of L-T4 therapy while simultaneously blocking the activity of the type-1 deiodinase with propylthiouracil (PTU).

Twenty hypothyroid patients who underwent total thyroidectomy or are affected by hypothyroidism and are on L-T4 therapy with normal TSH values will be recruited. After enrollment in the study, the patients eligibility will be determined during an outpatient visit. Patients will be admitted to the NIH Clinical Center for a 9-day period and will receive PTU at a dose of 200 mg four times daily for seven days. During the hospitalization for this research protocol, the following studies will be performed: serial blood sampling for circulating thyroid hormones to obtain pharmacokinetic parameters of T3, lipids, glucose and insulin; body composition; resting energy expenditure at room temperature and during exposure to mild cold; echocardiogram and EKG; skeletal muscle strength measurement and cardiac MRI.

The results obtained from this study will help in further characterizing the effects of thyroid hormone on metabolism, and may lead to important information on how to optimize the thyroid hormone replacement therapy for the treatment of hypothyroidism.

ELIGIBILITY:
* PARTICIPANT INCLUSION CRITERIA:

Study subjects will be adults older than 18 years who do not have any endogenous thyroid hormone production (i.e. status post total thyroidectomy, or in individuals who have a residual remnant greater than 2 mL, an uptake in the thyroid gland less than 5% while on therapy on 123I uptake scan) and on L-T4 replacement at a minimum dose of 1.6 microg/Kg in a steady state of euthyroidism.

EXCLUSION CRITERIA:

1. <TAB>Thyroid uptake > 5% at 24 hours on (123)I thyroid scan while on replacement therapy (in patients with thyroid gland residue > 2 mL by ultrasound).
2. <TAB>Patients who have lipid disorders requiring pharmacologic intervention.
3. <TAB>Any elevation of AST or ALT above upper limit of normal range.
4. <TAB>Any reduction of the WBC count below the lower limit of normal range.
5. <TAB>History of, and/or current diabetes mellitus (fasting glucose >126 mg/dL or current pharmacologic treatment).
6. <TAB>Hypertension requiring pharmacologic intervention.
7. <TAB>Female patients who are on hormonal contraceptives or are breastfeeding.
8. <TAB>Use of beta blocker medications and amiodarone.
9. <TAB>Pregnancy (women of child-bearing age must have a negative pregnancy test prior to inclusion).
10. <TAB>History of vasculitis, viral hepatitis (except A), granulocytopenia.
11. <TAB>Known allergy or serious adverse event to PTU.
12. <TAB>Current use of prescription medication or certain non-prescription medications and dietary supplements known to affect thyroid function and/or metabolism, or alter the pharmacokinetics of PTU. Should study volunteers receive other pharmacologic interventions a clinical pharmacist will be consulted to evaluate potential drug-drug interactions.
13. <TAB>Presence of persistent diarrhea or malabsorption syndromes that would interfere with the patient s ability to adequately absorb medications.
14. <TAB>Inability to obtain venous access for sample collection, or basal hemoglobin of less than or equal to 12 g/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01-04; Primary Completion 2013-11-29 (Actual); Study Completion 2013-11-29 (Actual)

PRIMARY OUTCOMES:
To assess the changes in glucose metabolism (hepatic gluconeogenesis and insulin-mediated glucose disposal). | 9 days
To serially evaluate the changes in end-organ effects of thyroid hormones during pharmacologic block of D1, specifically: 1. To assess the changes in lipid metabolism parameters (total cholesterol, LDL cholesterol, apolipoproteins). | 9 days
To assess the changes in resting energy expenditure. | 9 days
To assess the changes in facultative thermogenesis as measured in respiration chamber (at 19 (Infinite)C and 24 (Infinite)C). | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Francesco S Celi, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)

REFERENCES:
- [Background] Mentuccia D, Proietti-Pannunzi L, Tanner K, Bacci V, Pollin TI, Poehlman ET, Shuldiner AR, Celi FS. Association between a novel variant of the human type 2 deiodinase gene Thr92Ala and insulin resistance: evidence of interaction with the Trp64Arg variant of the beta-3-adrenergic receptor. Diabetes. 2002 Mar;51(3):880-3. doi: 10.2337/diabetes.51.3.880. PMID 11872697
- [Background] Mandel SJ, Berry MJ, Kieffer JD, Harney JW, Warne RL, Larsen PR. Cloning and in vitro expression of the human selenoprotein, type I iodothyronine deiodinase. J Clin Endocrinol Metab. 1992 Oct;75(4):1133-9. doi: 10.1210/jcem.75.4.1400883.
- [Background] Peeters RP, van Toor H, Klootwijk W, de Rijke YB, Kuiper GG, Uitterlinden AG, Visser TJ. Polymorphisms in thyroid hormone pathway genes are associated with plasma TSH and iodothyronine levels in healthy subjects. J Clin Endocrinol Metab. 2003 Jun;88(6):2880-8. doi: 10.1210/jc.2002-021592. PMID 12788902